CLINICAL TRIAL: NCT01510067
Title: Prevalence and Clinical Severity of Cutaneous Lupus Erythematosus
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Victoria Werth, Principal Investigator, University of Pennsylvania
Other Study IDs: 805758
Record Dates: First submitted 2012-01-10; First posted 2012-01-13 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Cutaneous Lupus Erythematosus (CLE)
Keywords: CLE; Lupus; Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Skin Tissue Biopsies
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The Cutaneous Lupus Erythematosus (CLE) database, established in 2006, is a multi-site database between the University of Pennsylvania and the University of Texas Southwestern (UTSW).

DETAILED DESCRIPTION:
The database has yielded valuable information and clinical insights into the pathophysiology, disease processes, treatments and quality of life associated with CLE. The CLE database incorporates the CLASI (Cutaneous Lupus Activity and Severity Index), a validated outcome measure of disease responsiveness in patients and other assessment tools, surveys and patient information to help validate the clinical course and quality of life of patients with CLE (cutaneous lupus erythematosus).

The CLE database has led to publication of significant studies on lupus and its clinical course, the effect of lupus on Quality of Life (QoL), including the effect of photosensitivity on QoL, and the effect of first line medications.

The CLE database is an ongoing resource that enables clinicians to evaluate the evolving clinical changes, treatment modalities and patient response to a challenging disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the criteria for having CLE, using the Gilliam classifications, and/or a diagnosis of systemic lupus erythematosus (SLE), using the American Rheumatism Association/American College of Rheumatology criteria. Subjects must be 18 years or older.

Exclusion Criteria:

* All subjects who do not meet the criteria for having CLE. Subjects who meet the criteria for CLE but who are not yet 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from among the patients seen at the Autoimmune Skin Disease Clinic at the Hospital of the University of Pennsylvania and other collaborating centers.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2006-12; Primary Completion 2030-01-02 (Estimated); Study Completion 2030-01-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Werth, M.D., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No